CLINICAL TRIAL: NCT06494033
Title: Prophylaxis Guided by Cytomegalovirus-specific T Cell Immunity to Prevent Cytomegalovirus Disease in Lung Transplant Recipients: a Single Center Prospective Study
Brief Title: Prophylaxis Guided by Cytomegalovirus-specific T Cell Immunity to Prevent Cytomegalovirus Disease in Lung Transplant Recipients
Status: Recruiting | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: Eurofins Viracor, LLC (Unknown)
Responsible Party: Principal Investigator, Yoichiro Natori, Associate Professor of Clinical, University of Miami
Other Study IDs: 20230432
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-12

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Prophylaxis guided by Cytomegalovirus-specific T cell Immunity: The immunological response of participants in this group will be followed for 1 year.

SUMMARY:
The purpose of this study is to evaluate the clinical outcomes of Cytomegalovirus (CMV) virus in the participants' body. Therefore, the study team will follow the participants' immunological response based on the Cytomegalovirus (CMV) virus testing.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients over 18 years of age
2. Lung transplant candidates with positive CMV IgG
3. Anticipated to receive a lung transplant (both double lung and single lung)

Exclusion Criteria:

1. Negative CMV IgG prior transplant
2. Pregnant or breastfeeding women
3. HIV infected patients
4. Combined organ (e.g., lung-heart, lung-kidney) transplant candidates

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants attending the Miami Transplant Institute.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Positive CMV Immunoglobulin (IgG) positive lung transplant | Up to 1 year
  Positive CMV Immunoglobulin (IgG) measured by IU/ml

SECONDARY OUTCOMES:
Graft Outcome status | Up to 1 year
  Graft Outcome status measured by number of rejection based on forced expiratory volume in 1 second( FEV1) /Forced vital capacity (FVC) ratio. A calculated ratio that helps diagnose obstructive and restrictive lung diseases
Number of dead participants | Up to 1 year
  Number of dead participants measured by numbers of death
Duration of CMV medication | Up to 1 year
  Duration of CMV medication measured by treatment days
Number of patients with CMV-positive results | Up to 1 year
  CMV disease measured by the number of patients with CMV-positive results
Severity of CMV Disease | Up to 1 year
  Severity of CMV disease measured by CMV polymerase chain reaction (PCR) (IU/mL)
Severity of Torque Teno virus | Up to 1 year
  Severity of Torque Teno virus measured by Torque Teno virus (TTV) (BAU/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Yoichiro Natori, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No